CLINICAL TRIAL: NCT04526678
Title: Iron Intake, Iron Status, Intestinal Health and Endurance Performance - Effects of Iron Supplementation in Young Female Football Players - a Pilot Study
Brief Title: Oslo Footballplayers Iron Supplementation and Training (FIT) Study
Acronym: Oslo-FIT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Life Sciences (Other)
Collaborators: Norwegian School of Sport Sciences (Other); University of Oslo (Other); Norwegian Olympic Sports Centre (Unknown)
Responsible Party: Principal Investigator, Siv K Bohn, Professor, Norwegian University of Life Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 969159570_KBM_SKB2020
Record Dates: First submitted 2020-08-13; First posted 2020-08-26 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Athletes; Iron; Endurance Performance; Hemoglobin; Intestinal Health; Microbiota
Keywords: oxidative stress; football
MeSH Terms: interventions — Iron-Dextran Complex

STUDY DESIGN:
Intervention Model Description: The intervention group will ingest 27 mg iron supplement per day for three months while the control group will not ingest iron supplements.
Who Masked: Outcomes Assessor
Masking Description: The assessor of outcomes are blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Iron supplements (Experimental): The intervention group will ingest 27 mg iron supplement per day for three months while the control group will not ingest iron supplements.
  Interventions: Dietary Supplement: Iron supplement (27mg)
- Control group (No Intervention): The control group will not ingest iron supplements.

INTERVENTIONS:
Dietary Supplement: Iron supplement (27mg) — The participants will be randomized to an intervention group or a control group. The intervention group will ingest 27mg iron daily for three months.
  Arms: Iron supplements

SUMMARY:
The aim of the study is to characterize the diet and iron status of young female elite football players and examine the relationship between iron intake, iron status, hemoglobin levels, intestinal health and sports performance. In addition, the effects of low-dose iron supplements on iron stores will be investigated and whether such supplementation affects intestinal health, microbiota composition and biomarkers for oxidative stress.

DETAILED DESCRIPTION:
Iron deficiency can lead to fatigue and anemia. Because iron is necessary for the formation of new blood cells (hematopoiesis), it is an extensive practice internationally among athletes to take iron supplements in the belief that this will improve endurance performance and oxygen transport capacity by increasing red blood cell production. Although iron intake in menstruating women has shown to reduce the prevalence of anemia and iron deficiency as well as increasing hemoglobin values and iron stores. However iron supplementation increases the risk of iron excess and can result in undesirable effects such as constipation and abdominal pain as well as negative impact on intestinal epithelial permeability and increase in oxidative stress. Because iron is important for the replication and survival of almost all bacteria, with few exceptions, the intake of iron also affect the composition of the intestinal bacteria. Not surprisingly, both high and low iron levels affect the composition of the microbiota in the gut.

It is not known if young menstruating Norwegian female athletes cover their need for iron via the diet or whether extra intake in the form of a low-dose supplement could be beneficial in terms of hemoglobin levels and sports performance. Because iron preparations are not prescription and are sold in pharmacies, health food stores and larger grocery stores, this can lead to uncritical intake of iron. Since the use of iron preparations has been documented to be widespread in foreign sports environments, it is important to both characterize the iron status of Norwegian athletes and at the same time examine the beneficial value of iron supplements on sports performance as well as monitoring effects on microbiota composition and intestinal health.

The aim of the study is therefore to characterize the diet and iron status of young female elite football players and examine the relationship between iron intake, iron status, hemoglobin levels, intestinal health and sports performance. In addition, the effects of low-dose iron supplements will be investigated in relation to iron stores, hemoglobin levels and sports performance and whether such supplementation affects intestinal health, microbiota composition and biomarkers for oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

- Female elite football players from two selected football clubs

Exclusion Criteria:

* Pregnancy
* Medical conditions that are worsened by taking iron supplements
* Already taking iron supplements

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Invited female elite football players from two selected football clubs.
Enrollment: 26 (Estimated)
Dates: Start 2020-08-11 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Diet composition | 3 months
  Diet composition will be assessed using digital 7 day dietary records.
Iron intake | 3 months
  Iron intake will be calculated based on average daily intake of iron according to the digital 7 day dietary recordings.
Serum Iron | 3 months
  Iron status will be assessed by analyzing serum iron (µmol/L)
Serum transferrin | 3 months
  Iron status will be assessed by analyzing serum transferrin (µmol/L)
Serum ferritin | 3 months
  Iron status will be assessed by analyzing serum ferritin (µg/L)
Hemoglobin levels | 3 months
  hemoglobin (Hb) (g/dl) will be analyzed in whole blood (EDTA) using an automated hematology analyzer.
LPS binding protein | 3 months
  -Intestinal health will be measured using biomarkers of intestinal leakage in serum and feces such as sLPS binding protein (LBP) (ug/ml)
Neutrophil gelatinase-associated lipocalin | 3 months
  -Intestinal health will be measured using biomarkers of intestinal leakage in serum and feces such as fecal neutrophil gelatinase-associated lipocalin (NGAL) (ng/g feces)
Serum cytokines | 3 months
  -Intestinal health will be measured using serum biomarkers of systemic inflammation (e.g. serum cytokines such as IL-1, IL-6, and TNF-α pg/ml).
Sports performance | 3 months
  Sports performance specific for football will be be measured using the Yo-Yo Intermittent Recovery Test (YYIR1).
Differential counts | 3 months
  Differential counts (% of WBC) will be analyzed in whole blood (EDTA) using an automated hematology analyzer.
Ferric reducing ability of plasma | 3 months
  -Oxidative stress will be assessed measuring the ferric reducing ability of plasma (FRAP)
Diacron reactive oxygen metabolites | 3 months
  -Oxidative stress will be assessed measuring biomarkers of total oksidativ stress e.g. diacron reactive oxygen metabolites (dROM).
Microbiota composition | 3 months
  -Microbiota composition will be analyzed mainly using 16S rRNA gene sequencing. The main effect of the intervention on the microbiota will be tested based on crude alpha and beta diversity indices but we will also apply advanced multivariate methods.

CONTACTS AND LOCATIONS:
Locations (1):
- Norwegian University of Life Sciences, Ås, Norway

IPD SHARING:
Plan to Share IPD: Undecided
An IPD sharing plan is not ready for the project